CLINICAL TRIAL: NCT00808704
Title: Effect of Erythropoietin on Neonatal Hypoxic Ischemic Encephalopathy
Brief Title: Neurological Outcome After Erythropoietin Treatment for Neonatal Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Collaborators: Zhengzhou Children's Hospital, China (Other); Medical University Innsbruck (Other); Göteborg University (Other)
Responsible Party: Professor Xiaoyang Wang, Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HN-200312
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: asphyxia; erythropoietin; neonates
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: recombinant human erythropoietin — r-hu-EPO were administered either 300 U/kg or 500 U/kg, subcutaneously the first time and then intravenously every other day for 2 weeks.
  Other Names: EPO

SUMMARY:
Perinatal asphyxia-induced brain injury is one of the most common causes of morbidity and mortality in term and preterm neonates, accounting for 23% of neonatal deaths globally. Although many neuroprotective strategies appeared promising in animal models, most of them have failed clinically. Erythropoietin (EPO) is an endogenous cytokine originally identified for its role in erythropoiesis. Clinical trial has demonstrated the safety and efficacy of recombinant human erythropoietin (r-hu-EPO) in the prevention or treatment of anemia of prematurity. To date, there are no reports evaluating possible effects of EPO on neonatal HIE.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy of the newborn infant remains a significant socio-economic health problem worldwide. Moderate to severe HIE of newborn infants is associated with a high rate of death or long-term disabilities. Historically, treatment has been purely supportive including stabilizing cardio-respiratory functions and treating convulsions.Recent multi-center trials assessing the effects of hypothermia demonstrated improved outcome in term neonates with moderate hypoxic-ischemic encephalopathy (HIE). However, hypothermia was not effective beyond 6 hrs after brain injury.

Systemically administered EPO was neuroprotective in neonatal brain injury models. Clinical study on adult stroke showed improved outcome. However, treating HIE with EPO raises a series of questions such as: i) Can the patient population of this study readily be compared with those in the hypothermia trials? ii) What are the pharmacokinetics of EPO, including issues of dosage and timing, and does administered EPO cross the blood-brain-barrier? iii) How does the effectiveness, side effects and potentials of EPO therapy compare with induced hypothermia?

ELIGIBILITY:
Inclusion Criteria:

* Apgar score of 5 or less at 5 min after birth or continued need for resuscitation, including endotracheal or mask ventilation at 10 min after birth.
* The severity of encephalopathy, moderate or severe, was assessed by certified examiners according to the criteria of Sarnat and Sarnat(13), consisting of altered state of consciousness: lethargy, stupor or coma, and at least one or more of hypotonia, abnormal reflexes including oculomotor or pupillary abnormalities, absent or weak sucking or clinical seizures.

Exclusion Criteria:

* Major congenital abnormalities, head trauma or skull fracture causing major intracranial hemorrhage, mild HIE, financial problems of the parents, lack of permanent address or postnatal age > 48 hrs

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Mortality and disability rate. Mortality and disability rate at 18months of age. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Changlian Zhu, MD, PhD, Study Director — Zhengzhou University
Locations (1):
- NICU, the Third Affiliated Hospital, Zhengzhou University, Zhengzhou, Henan, China